CLINICAL TRIAL: NCT05031442
Title: A Randomized Study of Pant Type Absorbing Urinary Incontinence Products With Cross-over Design
Brief Title: Study of Pant Type Absorbing Urinary Incontinence Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essity Hygiene and Health AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R-ONE
Record Dates: First submitted 2021-08-11; First posted 2021-09-01 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Subjects use one product for 5 days and then switch to another product for 5 days. One of the products is the investigational product and one is the reference product.
Masking Description: Participants are randomized to start with either reference or investigational product. The type of product is masked for the participant but since there are slight differences between the products the masking cannot be ensured.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- low waist arm (investigational product RH1 first) (Other): Investigational product RH1 (low waist) will be used for 5 consecutive days at the start before switching to the control product (low waist) for 5 days after cross-over.
  Interventions: Device: RH1 (low waist); Device: Reference variant 1 (low waist)
- high waist arm (Investigational product RC2 first) (Other): Investigational product RC2 (high waist) to be used for 5 consecutive days at the start before switching to the control product (high waist) for 5 days after cross-over.
  Interventions: Device: RC2 (high waist); Device: Reference variant 2 (high waist)
- low waist arm (Control product first) (Other): Control product (low waist) to be used for 5 consecutive days at the start before switching to the investigational product RH1 for 5 days after cross-over.
  Interventions: Device: RH1 (low waist); Device: Reference variant 1 (low waist)
- high waist (Control product first) (Other): Control product (high waist) to be used for 5 consecutive days at the start before switching to the investigational product RC2 for 5 days after cross-over.
  Interventions: Device: RC2 (high waist); Device: Reference variant 2 (high waist)

INTERVENTIONS:
Device: RH1 (low waist) — Investigational product variant 1 low waist
  Arms: low waist arm (Control product first); low waist arm (investigational product RH1 first)
Device: Reference variant 1 (low waist) — Reference product variant 1
  Other Names: TENA Silhouette Normal Low waist
  Arms: low waist arm (Control product first); low waist arm (investigational product RH1 first)
Device: RC2 (high waist) — Investigational product variant 2 high waist
  Arms: high waist (Control product first); high waist arm (Investigational product RC2 first)
Device: Reference variant 2 (high waist) — Reference product variant 2
  Other Names: TENA Silhouette Normal High waist
  Arms: high waist (Control product first); high waist arm (Investigational product RC2 first)

SUMMARY:
Pre-market feasibility clinical investigation designed to evaluate the clinical performance and safety of the investigational product in its intended target population

DETAILED DESCRIPTION:
The clinical clinical investigation is prospective, cross-over, interventional, multicentre and pre-market. The investigation aims to demonstrate the performance and safety of a new absorbing hygiene product (medical device) when used as intended in subjects affected with light to medium urinary incontinence compared to a reference (control) product representing standard of care.

The study participants will be randomly assigned to one of 4 groups. Each group will receive a predefined pair of investigational and reference products (variants: either high waist or low waist) to be used in a predefined order (crossover design: investigational or reference product to be used first). Hence, each study subject will use two products (one investigational product and a corresponding reference product of the same variant) and act as its own control. The study subjects will use one product for 5 days and then switch to use the other product for 5 days.

The primary endpoint for the investigation is the comparison in leakage performance of the investigation product with the reference product. There are also secondary endpoints regarding safety and product satisfaction and product preference.

ELIGIBILITY:
Inclusion Criteria:

* Adult women between age 45 and 75.
* Be willing and able to provide informed consent.
* Capability and willingness to follow the protocol.
* Experience incontinence daily or at least two times a week.
* Uses some sort of protection for the incontinence daily or at least two times a week.
* Uses five or more pieces of protection per week.
* Is currently using protective underwear; a pull-up (pant) product made for incontinence.
* Is able to wear a pant product of size M.
* Is currently using TENA Silhouette or Always Discreet Boutique product.
* Should be affiliate to the social security system.

Exclusion Criteria:

* Is pregnant or nursing.
* Known allergies or intolerances to one or several components of the investigational products.
* Be dependent on either alcohol or recreational drugs.
* Participation in an investigational study of a drug, biologic, or device within 30 days prior to entering the clinical investigation or planned during the course of the clinical investigation.
* Being under safeguard and protection of justice
* Having cognitive impairments.
* Any other condition that may make participation in the clinical investigation inappropriate, as judged by investigator.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Diary reported number of urinary leakages | Through study completion until Day 12 +/-2
  The proportion of products experiencing urine leakage over the 5 day test period is compared between the investigational and reference product. A diary is used to collect this information for each used product.

SECONDARY OUTCOMES:
Incidence of safety events | Through study completion until Day 12 +/-2
  The number and severity of reported safety events are collected and compared for the intervention and reference products.
Product satisfaction questionnaire | Day 6 +/-1
  Overall satisfaction score with investigational product as compared to the reference product using a 5-point likert scale.
Product satisfaction questionnaire | Day 12 +/-2
  Overall satisfaction score with investigational product as compared to the reference product using a 5-point likert scale.
Product preference questionnaire | Measured on day 12 +/-2
  Subject preference score for the investigational product as compared to the reference product using a 5-point likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Paquet Labertrande, MD, Principal Investigator
Locations (3):
- France (3):
  - Eurofins Optimed, Gières
  - Intertek, Paris
  - LyREC, Pierre-Bénite